CLINICAL TRIAL: NCT04198779
Title: Interest of the Smartphone Application "MonCœur" in the Follow-up of Patients With Heart Failure
Acronym: APPLIMONCOEUR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recrutement rate
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-01
Record Dates: First submitted 2019-12-06; First posted 2019-12-13 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Heart Decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, randomized, controlled, open, 2 parallel arms study, in 11 centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APPLI (Experimental): Care support with implementation of the application
  Interventions: Device: APPLI
- CONTROL (No Intervention): Conventional care support

INTERVENTIONS:
Device: APPLI — The support with the digital application is including a 10-minutes training about the use of the digital application at the beginning of the study. Patient will have to register information about their Heart failure disease (weight, shortness of breath, fatigue, mood, cardiologist appointments, blood results, ...). During each routine consultation, patients will be encouraged to use the digital app, and the obstacles encountered will be explored and resolved. In addition, participants will receive an email containing relevant information and, every three months, an email reminder of the use of the application.
  Arms: APPLI

SUMMARY:
Heart failure is a chronic disease that requires careful monitoring and therapeutic education. Smartphones have made their appearance in patients lives and allow close contact with them. The possibility of using a digital application dedicated to patients with heart failure concerning the symptoms to be monitored, treatments, diet, appointments, physical activity could improve the monitoring and the prognosis of patients following their hospitalization.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate that the use of a special application dedicated to the monitoring of heart failures disease has a favorable impact on the occurrence of readmissions and, ultimately, cardiovascular mortality. The aim of this study is also to demonstrate that the use of this "MonCœur" application improves symptoms, quality of life, treatment compliance, diet compliance, and physical activity in patient with heart failure disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for acute or decompensated heart failure
* Patient with a smartphone and able to use a digital application
* Beneficiary of a social protection scheme
* Patients benefiting from a telemedicine program can be included

Exclusion Criteria:

* Acute coronary syndrome during ongoing hospitalization.
* Acute myocarditis, constrictive pericarditis, acute endocarditis during ongoing hospitalization.
* Isolated right heart failure of respiratory origin.
* Existence of a cause considered rapidly reversible to acute heart failure: tachyarrhythmia, excessive bradycardia, acute anemia, acute renal failure, malignant hypertension, overdose or cardiotoxic drug intoxication.
* Indication of cardiac surgery scheduled within 3 months after hospitalization, patients with Tavi or MItraclip expected within 3 months
* Extracardiac disease with short-term prognosis (progressive neoplasia).
* Refusal or incapacitation of language or psychic to sign informed consent
* Patients participating in an other biomedical research can not participate in this study for the first 6 months, not to interfere with the consultation process of the study.
* Pregnant or lactating women can't participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of the use of "MonCoeur" application on the impact of patient health self-care | 3, 6 and 12 months
  Comparison between the 2 study arms of the score of the European Heart Failure Self-care Behaviour Scale, consisting of 9 items each evaluated on a 5-point Likert scale, and allowing the calculation of a standardized global score from 0 to 100: the highest score indicating better "self-care".

SECONDARY OUTCOMES:
Evaluation of the use of "MonCoeur" application on hospitalisation rate | 3, 6 and 12 months
  Comparison between the 2 study arms on the number of days without hospitalisation
Evaluation of the use of "MonCoeur" application on cardiovascular parameters | 3, 6 and 12 months
  Comparison between the 2 study arms of Brain Natriuretic Peptid (nanograms / liter)
Evaluation of the use of "MonCoeur" application on patient compliance | 3, 6 and 12 months
  Comparison between the 2 study arms on percentage of appointments scheduled versus appointments honored. Comparison between the 2 study arms of the score of the treatment observance scale Ameli.
Evaluation of the use of "MonCoeur" application on patient quality of life: Minnesota Living with Heart Failure Questionnaire | 3, 6 and 12 months
  Comparison between the 2 study arms of the score of the Minnesota Living with Heart Failure Questionnaire. It provides a total score (range 0-105, from best to worst), as well as scores for two dimensions, physical (8 items, range 0-40) and emotional (5 items, range 0-25). The other eight items (of the total of 21) are only considered for the calculation of the total score.
Evaluation of the use of "MonCoeur" application on patient physical activity | 3, 6 and 12 months
  Comparison between the 2 study arms of the score of the Qappa ("questionnaire d'activité physique pour personnes âgées" / translation in english: "physical activity questionnaire for seniors") physical activity questionnaire. The QAPPA uses the calculation system of the volume of physical activity per minute and per week and classified as high, moderate, or low level.
Describe how often and how the application is used by patients | 3, 6 and 12 months
  Calculation of the number and type of parameters filled in the application.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle BERTHELOT, MD, Principal Investigator — Hôpital Bicêtre
Locations (16):
- France (16):
  - CHU Amiens - Picardie - Site Sud, Amiens
  - Hospices Civils de Lyon, Bron
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU de Lille, Lille
  - Groupe Hospitalier Sud Ile de France, Melun
  - CHU Arnaud de Villeneuve, Montpellier
  - Hôpital Lariboisière, Paris
  - Hôpital Universitaire Pitié Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU de Poitiers, Poitiers
  - CHU de ROUEN - Hôpital Charles Nicolle, Rouen
  - CHRU de Strasbourg, Strasbourg
  - Hôpital Sainte Musse de Toulon, Toulon
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No